CLINICAL TRIAL: NCT07292207
Title: Phase 2 Study of Abemaciclib for Molecular Residual Disease Detected by Circulating Tumor DNA in HR+/HER2- Early Breast Cancer
Brief Title: Abemaciclib for Molecular Residual Disease Detected by Circulating Tumor DNA in HR+/HER2- Early Breast Cancer
Acronym: ARCHE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nagoya City University (Other)
Collaborators: Tohoku University (Other); Japanese Foundation for Cancer Research (Other); National Cancer Center, Japan (Other Government); University of Tsukuba (Other); Gifu University Graduate School of Medicine (Other); Aichi Cancer Center (Other)
Responsible Party: Principal Investigator, Kazuki Nozawa, Principal Investigator, Nagoya City University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCU-003-Abema; NCU (Other: Nagoya City University)
Record Dates: First submitted 2025-11-22; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: ctDNA Monitoring; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib; Tablets

STUDY DESIGN:
Intervention Model Description: Abemaciclib for 2-year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment for MRD positive (Experimental): ctDNA-posotive during adjuvant treatment
  Interventions: Drug: Abemaciclib 150 MG Oral Tablet

INTERVENTIONS:
Drug: Abemaciclib 150 MG Oral Tablet — Adding abemaciclib for 2-year with endcrine treatment

SUMMARY:
The goal of this clinical study is to determine whether monitoring ctDNA and treating patients who become ctDNA-positive with abemaciclib can help prevent the recurrence of hormone receptor-positive, HER2-negative breast cancer after curative surgery and standard therapy. The study will also assess the safety of abemaciclib and the medical problems that may occur during treatment. Participants will receive routine follow-up after surgery, undergo regular blood tests to measure ctDNA, and, if ctDNA becomes positive, receive abemaciclib for a defined treatment period with scheduled clinic visits for examinations and safety assessments. Researchers will evaluate recurrence-free survival, distant recurrence-free survival, adverse events, the time between ctDNA positivity and clinical recurrence, and the rate of ctDNA clearance at the end of abemaciclib therapy.

DETAILED DESCRIPTION:
The purpose of this clinical study is to investigate whether identifying molecular relapse through ctDNA monitoring and initiating abemaciclib treatment at the time of ctDNA positivity can reduce the risk of recurrence in patients with hormone receptor-positive, HER2-negative early breast cancer who have completed curative surgery and standard adjuvant therapy. The study also aims to evaluate the safety profile of abemaciclib in this early-stage setting and to clarify how patients tolerate the treatment over time. Participants will undergo routine postoperative surveillance, including scheduled imaging and laboratory testing, as well as regular blood sampling for ctDNA analysis. When ctDNA becomes detectable, indicating minimal residual disease, participants will begin a predefined course of abemaciclib and attend clinic visits at regular intervals for physical examinations, toxicity assessments, and laboratory monitoring.

In addition to determining whether early intervention with abemaciclib can delay or prevent clinical recurrence, researchers will examine several key outcomes. These include invasive disease-free survival, distant recurrence-free survival, and the incidence of adverse events throughout the treatment period. The study will also measure the "lead time" between ctDNA positivity and radiologic or clinical recurrence, which may provide insight into the biological dynamics of disease relapse. Furthermore, researchers will evaluate ctDNA clearance at the completion of abemaciclib therapy, as ctDNA clearance may serve as an early indicator of treatment efficacy. Collectively, these results are expected to clarify the clinical utility of ctDNA-guided therapy escalation and to inform future strategies for preventing recurrence in early breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer.
* ctDNA-positive after completion of definitive local/systemic therapy.
* Definitive breast surgery performed; axillary node status confirmed.
* HR-positive, HER2-negative disease.
* Tumor and nodal status meet predefined pathological risk criteria.
* ECOG PS 0 - 1.
* No bilateral breast cancer.
* Adequate recovery from prior therapy and acceptable organ function.
* No distant metastasis before registration.
* Appropriate contraception; informed consent obtained.

Exclusion Criteria:

* Active second malignancy.
* Prior CDK4/6 inhibitor use.
* Recent major surgery or active infection.
* Uncontrolled hypertension or significant cardiac disease.
* Recent thromboembolic events.
* Interstitial lung disease or active pneumonitis.
* Unrecovered toxicities from prior treatment.
* Active HIV, HBV, or HCV infection.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2031-08-31 (Estimated)

PRIMARY OUTCOMES:
ctDNA clearance rate | Within 2 years
  The rate of change of ctDNA positive to negative during abemaciclib treatment

SECONDARY OUTCOMES:
Invasive disease-free survival (IDFS) | through study completion, an average of 3 year
  A measure of the time from study enrollment until any invasive recurrence, second primary cancer, or death occurs.
Distant recurrence-free survival (DRFS) | through study completion, an average of 3 year
  The time from study enrollment to the development of distant metastatic recurrence or death.
Lead time from ctDNA positivity to clinical recurrence | through study completion, an average of 2 year
  The interval between the first detection of ctDNA positivity and the confirmed clinical or radiologic recurrence of cancer.
Incidence of adverse events | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ryuta Asada, PhD, Study Director — Nagoya City University
Locations (1):
- Nagoya City University, Nagoya, Japan

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol
Time Frame: 1 year after publication.
Access Criteria: All researcher